CLINICAL TRIAL: NCT01536587
Title: Effects of Bronchodilatation With Salmeterol on the Autonomic Nervous System
Brief Title: Effects of Salmeterol on Autonomic Nervous System
Acronym: ESAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 114520
Record Dates: First submitted 2012-02-02; First posted 2012-02-22 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: influence of bronchodilatation with salmeterol on the autonomic nervous systems in COPD patients will be measured using MSNA.; Relation of COPD and sympathetic nerve activity is to be evaluated,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): Inhalation of salmeterol 50 µg twice daily over 4 weeks
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: Salmeterol — At visit 1 the sympathetic activity will be registered using microneurographic recordings of efferent muscle sympathetic nerve activity (MSNA) in the peroneal nerve and respiration over 2 hours, after 20 minutes of recording, 1 dose of placebo will be administered and after a further recording period of 45 minutes a dose of salmeterol 50 µg will be administered which will be followed by a further period of data registration. At visit 2 following 4 weeks of inhaled treatment with salmeterol the same procedures will be performed but a placebo inhalation will not be performed.

SUMMARY:
This is a 4-week non-randomized, partially blinded, single-arm monocentre study in subjects with Chronic Obstructive Pulmonary Disease (COPD) Global Initiative for Chronic Obstructive Lung Disease (GOLD) class II or III with the aim to demonstrate that inhaled therapy with salmeterol reduces sympathetic activity as evaluated by microneurography. A maximum of 32 subjects is planned to be enrolled.

DETAILED DESCRIPTION:
This is a 4-week non-randomized, partially blinded, single-arm monocentre study in subjects with COPD GOLD class II or III with the aim to demonstrate that inhaled therapy with salmeterol reduces sympathetic activity as evaluated by microneurography. A maximum of 32 subjects is planned to be enrolled.

During a complex data registration period comprising the continuous recording of muscle sympathetic nerve activity (MSNA) and respiration and of various other measurements at Visit 1, placebo and 50 μg of salmeterol via Diskus™ inhaler will be administered in a sequential design. Following Visit 1, the subjects will be treated with salmeterol 50 μg twice daily via Diskus inhaler for 4 weeks. At the Final Visit (Visit 2) the data registration period of Visit 1 will be repeated with the only difference that no placebo will be administered.

Further endpoints, besides the evaluation of MSNA, include heart rate variability (HRV), spontaneous baroreflex sensitivity and lung function parameters.

Study enrolment will be stopped when valid MSNA data on the immediate effect of inhalation (manoeuvres at Visit 1) are available for 24 subjects.

ELIGIBILITY:
Inclusion Criteria:

* COPD of GOLD Class II or III with a post-bronchodilator spirometry forced expiratory volume in one second (FEV1) <60% predicted and FEV1/vital capacity (VC) <70% in accordance with the GOLD executive summary
* Subject is ambulatory (outpatient)
* Subject is therapy-naive (defined as not receiving any previous regular COPD therapy)
* Subjects with a current or prior history of ≥10 pack-years of cigarette smoking at Screening Visit. Previous smokers are defined as those who have stopped smoking for at least 1 month prior to Visit 1
* Willing to participate in the study, must be able to inhale study medication

Exclusion Criteria:

* Women who are pregnant or lactating
* Subjects not willing or unable to sign the informed consent before study start
* diagnosis of asthma
* α-1 antitrypsin deficiency
* active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases
* Subjects with lung volume reduction surgery within the 12 months prior to Screening
* Subjects who have been hospitalized due to poorly controlled COPD within 6 weeks prior to the Screening Visit
* Subjects with poorly controlled COPD, defined as the occurrence of an exacerbation managed with systemic corticosteroids or antibiotics prescribed by a physician 6 weeks prior to the Screening Visit
* Frequent exacerbations necessitating the therapy with inhaled glucocorticosteroids according to the GOLD guideline
* COPD with nasal intermittent positive pressure ventilation (NIPPV)
* Treatment with drugs having direct sympathomimetic activity (e.g. theophylline, moxonidine, clonidine), Oral medication with beta2-sympathomimetics
* Inhaled therapy with anti-cholinergics, sodium cromoglycate or nedocromil sodium
* Treatment with systemic, oral or parenteral (intra-articular) corticosteroids
* Treatment with strong cytochrome P450 3A4 inhibitors
* Treatment with any other investigational drug
* Oxygen therapy: Subjects receiving treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day
* Subjects who are medically unable to withhold their short-acting beta-agonist (SABA) for the 6-hour period required prior to spirometry testing at each study visit
* Subjects with clinically significant sleep apnoea that is uncontrolled
* Unstable angina pectoris or signs and history of left heart failure with a left ventricular ejection fraction <40%
* Arterial hypertension necessitating treatment with >1 antihypertensive drug
* Clinically evident polyneuropathy
* Diabetes mellitus necessitating any pharmacological therapy
* Severe concomitant disease (likely to reduce life expectancy to less than 3 years)
* Other diseases/abnormalities: Subjects with historical or current evidence of clinically significant neurological, psychiatric, renal, hepatic, immunological, endocrine or haematological abnormality that is uncontrolled

Ages: 41 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Göttingen, Lower Saxony, Germany

REFERENCES:
- [Derived] Haarmann H, Mohrlang C, Tschiesner U, Rubin DB, Bornemann T, Ruter K, Bonev S, Raupach T, Hasenfuss G, Andreas S. Inhaled beta-agonist does not modify sympathetic activity in patients with COPD. BMC Pulm Med. 2015 Apr 30;15:46. doi: 10.1186/s12890-015-0054-7. PMID 25924990

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Visit 1, a complex data registration was performed during which placebo and 50 micrograms (µg) salmeterol via SEREVENT DISKUS inhaler was administered sequentially. Following Visit 1, participants were treated with salmeterol 50 µg twice daily (BID) via DISKUS inhaler for 4 weeks.
Groups:
- Salmeterol 50 µg BID: Participants received salmeterol 50 micrograms (µg) via DISKUS inhaler twice daily (BID) over the course of 4 weeks.
Period: Overall Study
Arm/Group | Salmeterol 50 µg BID
Started | 32
Completed | 30
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.19 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Muscle Sympathetic Nerve Activity (MSNA) at 2 Hours (Week 0)
Description: Human MSNA is composed of vasoconstrictor impulses grouped in pulse synchronous bursts that usually occur in sequences, preferentially during transient reductions of blood pressure. Sympathetic activity was measured using microneurographic recordings of efferent in the peroneal nerve. MSNA reflects sympathetic discharge to the vascular bed of the skeletal muscle. The change in MSNA (bursts per 100 heart beats [bursts/100 heart beats]) was calculated as the difference in MSNA change from Baseline to after the inhalation of salmeterol (2 hours, Week 0, Visit 1) minus the MSNA change from Baseline to after the inhalation of placebo (1 hour, Week 0, Visit 1).
Time Frame: Baseline and 2 hours (Week 0)
Population: ITT-MSNA Population: all participants who received at least one dose of study medication and who had a valid data registration period of the primary endpoint.
Measure: Mean (Standard Deviation); unit: Bursts/100 heart beats
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 18
Bursts/100 heart beats | -1.3 (8.13)
Statistical Analysis 1: Comparison: Salmeterol 50 µg BID; Test type: Superiority or Other; p = 0.5062, paired t-Test, 2-sided

2. Secondary Outcome: Change From Baseline in MSNA (Evaluated by Microneurography as Bursts/100 Heart Beats) at Week 4
Description: Human MSNA is composed of vasoconstrictor impulses grouped in pulse synchronous bursts that usually occur in sequences, preferentially during transient reductions of blood pressure. Sympathetic activity was measured using microneurographic recordings of efferent in the peroneal nerve. MSNA reflects sympathetic discharge to the vascular bed of the skeletal muscle. Change in MSNA is expressed in terms of bursts per 100 heart beats (bursts/100 heart beats). Change from Baseline was calculated as the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline and Week 4
Population: ITT-MSNA Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Bursts/100 heart beats
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 12
Bursts/100 heart beats | -3.1 (11.58)

3. Secondary Outcome: Change From Baseline in MSNA (Evaluated by Microneurography as Bursts/Minute) at 2 Hours (Week 0)
Description: Human MSNA is composed of vasoconstrictor impulses grouped in pulse synchronous bursts that usually occur in sequences, preferentially during transient reductions of blood pressure. Sympathetic activity was measured using microneurographic recordings of efferent in the peroneal nerve. MSNA reflects sympathetic discharge to the vascular bed of the skeletal muscle. The change in MSNA (bursts per minute [bursts/minute]) was calculated as the difference in MSNA change from Baseline to after the inhalation of salmeterol (2 hours, Week 0, Visit 1) minus the MSNA change from Baseline to after the inhalation of placebo (1 hour, Week 0, Visit 1).
Time Frame: Baseline and 2 hours (Week 0)
Population: ITT-MSNA Population
Measure: Mean (Standard Deviation); unit: Bursts/minute
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 18
Bursts/minute | 0.3 (5.60)

4. Secondary Outcome: Change From Baseline in MSNA (Evaluated by Microneurography as Bursts/Minute) at Week 4
Description: Human MSNA is composed of vasoconstrictor impulses grouped in pulse synchronous bursts that usually occur in sequences, preferentially during transient reductions of blood pressure. Sympathetic activity was measured using microneurographic recordings of efferent in the peroneal nerve. MSNA reflects sympathetic discharge to the vascular bed of the skeletal muscle. Change in MSNA is expressed in terms of bursts per minute (bursts/minute). Change from Baseline was calculated as the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline and Week 4
Population: ITT-MSNA Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Bursts/minute
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 12
Bursts/minute | 0.5 (7.58)

5. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Standard Deviation of NN Intervals (SDNN) at 2 Hours (Week 0) and at Week 4 (ITT Population)
Description: Heart rate variability (HRV) refers to the complex beat-to-beat (NN) variation in heart rate produced by the interplay of sympathetic and parasympathetic neural activity at the sinus node of the heart. SDNN reflects all the cyclic components responsible for variability in the period of recording; therefore, it represents total variability. Change in HRV (SDNN) after salmeterol inhalation is expressed in terms of milliseconds (ms). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
ms
  Change from Baseline to 2 hours, Week 0, n=32 | -1.7 (26.4)
  Change from Baseline to Week 4, n=31 | 0.1 (53.9)

6. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Standard Deviation of NN Intervals (SDNN) at 2 Hours (Week 0) and at Week 4 (ITT-MSNA Population)
Description: HRV refers to the complex beat-to-beat (NN) variation in heart rate produced by the interplay of sympathetic and parasympathetic neural activity at the sinus node of the heart. SDNN reflects all the cyclic components responsible for variability in the period of recording; therefore, it represents total variability. Change in HRV (SDNN) after salmeterol inhalation is expressed in terms of milliseconds (ms). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT-MSNA Population
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 18
ms
  Change from Baseline to 2 hours, Week 0 | 1.2 (22.5)
  Change from Baseline to Week 4 | -12.1 (29.5)

7. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Square Root of the Mean Squared Difference of Successive NNs (RMSSD) at 2 Hours (Week 0) and at Week 4 (ITT Population)
Description: HRV refers to the complex beat-to-beat (NN) variation in heart rate produced by the interplay of sympathetic and parasympathetic neural activity at the sinus node of the heart. Compared with SDNN, RMSSD is a short-term variation of heart rate. Change in HRV (RMSSD) after salmeterol inhalation is expressed in terms of milliseconds (ms). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
ms
  Change from Baseline to 2 hours, Week 0, n=32 | -11.5 (36.3)
  Change from Baseline to Week 4, n=31 | -5.2 (96.1)

8. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Square Root of the Mean Squared Difference of Successive NNs (RMSSD) at 2 Hours (Week 0) and at Week 4 (ITT-MSNA Population)
Description: as for outcome 7
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT-MSNA Population
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 18
ms
  Change from Baseline to 2 hours, Week 0 | -10.6 (26.4)
  Change from Baseline to Week 4 | -32.5 (47.4)

9. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Absolute Low Frequency (LF) Power at 2 Hours (Week 0) and at Week 4 (ITT Population)
Description: HRV refers to the complex beat-to-beat (NN) variation in heart rate produced by the interplay of sympathetic and parasympathetic neural activity at the sinus node of the heart. HRV frequencies can be analyzed with frequency domain methods: the LF component of the HRV spectrum reflects sympathetic activity. Change in HRV (absolute LF) after salmeterol inhalation is expressed in terms of milliseconds squared (ms^2). Change from Baseline were calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
ms^2
  Change from Baseline to 2 hours, Week 0, n=32 | -123.8 (1588.4)
  Change from Baseline to Week 4, n=31 | -390.1 (1463.3)

10. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Absolute Low Frequency (LF) Power at 2 Hours (Week 0) and at Week 4 (ITT-MSNA Population)
Description: HRV refers to the complex beat-to-beat (N-N) variation in heart rate produced by the interplay of sympathetic and parasympathetic neural activity at the sinus node of the heart. HRV frequencies can be analyzed with frequency domain methods: The LF component of the HRV spectrum reflects sympathetic activity. Change in HRV (absolute LF) after salmeterol inhalation is expressed in terms of milliseconds squared (ms2). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation), respectively.
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT-MSNA Population
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 18
ms^2
  Change from Baseline to 2 hours, Week 0 | 220.7 (1038.2)
  Change from Baseline to Week 4 | -248.1 (755.2)

11. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Absolute High Frequency (HF) Power at 2 Hours (Week 0) and at Week 4 (ITT Population)
Description: HRV refers to the complex beat-to-beat (NN) variation in heart rate produced by the interplay of sympathetic and parasympathetic neural activity at the sinus node of the heart. HRV frequencies can be analyzed with frequency domain methods: the HF component of the HRV spectrum reflects parasympathetic activity. Change in HRV (absolute HF) after salmeterol inhalation is expressed in terms of milliseconds squared (ms^2). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
ms^2
  Change from Baseline to 2 hours, Week 0, n=32 | -457.9 (1591.6)
  Change from Baseline to Week 4, n=31 | 817.5 (8754.6)

12. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Absolute High Frequency (HF) Power at 2 Hours (Week 0) and at Week 4 (ITT-MSNA Population)
Description: as for outcome 11
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT-MSNA Population
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 18
ms^2
  Change from Baseline to 2 hours, Week 0 | -372.1 (1194.4)
  Change from Baseline to Week 4 | -840.2 (1491.5)

13. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Normalized Low Frequency (LF) Power at 2 Hours (Week 0) and at Week 4 (ITT Population)
Description: HRV refers to the complex beat-to-beat (NN) variation in heart rate produced by the interplay of sympathetic and parasympathetic neural activity at the sinus node of the heart. HRV frequencies can be analyzed with frequency domain methods: the LF component of the HRV spectrum reflects sympathetic activity. Change in HRV (normalized LF) after salmeterol inhalation is expressed in terms of normalized units that represent the relative value of LF power component in proportion to the total power minus the very LF (VLF) component (LF/(Total Power-VLF)*100). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
percent change
  Change from Baseline to 2 hours, Week 0, n=32 | 8.4 (14.5)
  Change from Baseline to Week 4, n=31 | 2.5 (23.3)

14. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Normalized Low Frequency (LF) Power at 2 Hours (Week 0) and at Week 4 (ITT-MSNA Population)
Description: as for outcome 13
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT-MSNA Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 18
percent change
  Change from Baseline to 2 hours, Week 0 | 10.8 (14.6)
  Change from Baseline to Week 4 | 11.6 (19.0)

15. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Normalized High Frequency (HF) Power at 2 Hours (Week 0) and at Week 4 (ITT Population)
Description: HRV refers to the complex beat-to-beat (NN) variation in heart rate produced by the interplay of sympathetic and parasympathetic neural activity at the sinus node of the heart. HRV frequencies can be analyzed with frequency domain methods: the HF component of the HRV spectrum reflects parasympathetic activity. Change in HRV (normalized HF) after salmeterol inhalation is expressed in terms of normalized units that represent the relative value of HF power component in proportion to the total power minus the very LF (VLF) component (HF/(Total Power-VLF)*100). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
percent change
  Change from Baseline to 2 hours, Week 0, n=32 | -8.4 (14.5)
  Change from Baseline to Week 4, n=31 | -2.5 (23.3)

16. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Normalized High Frequency Power (HF) at 2 Hours (Week 0) and at Week 4 (ITT-MSNA Population)
Description: as for outcome 15
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT-MSNA Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 18
percent change
  Change from Baseline to 2 hours, Week 0 | -10.8 (14.6)
  Change from Baseline to Week 4 | -11.6 (19.0)

17. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Heart Rate at 2 Hours (Week 0) and at Week 4 (ITT Population)
Description: Heart rate refers to the speed of the heartbeat, specifically the number of heartbeats per unit of time. Change in HRV (heart rate) after salmeterol inhalation is expressed in terms of the heart rate (beats) per minute (heart rate/min). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0 before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
beats per minute (bpm)
  Change from Baseline to 2 hours, Week 0, n=32 | 3.7 (4.2)
  Change from Baseline to Week 4, n=31 | 3.9 (4.3)

18. Secondary Outcome: Change From Baseline in Heart Rate Variability (HRV): Heart Rate at 2 Hours (Week 0) and at Week 4 (ITT-MSNA Population)
Description: as for outcome 17
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT-MSNA Population
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 18
beats per minute (bpm)
  Change from Baseline to 2 hours, Week 0 | 4.4 (4.7)
  Change from Baseline to Week 4 | 4.9 (4.8)

19. Secondary Outcome: Change From Baseline in Spontaneous Baroreflex Sensitivity (BRS) at 2 Hours (Week 0) and at Week 4 (ITT Population)
Description: BRS is an important characteristic of baroreflex control and is often noninvasively assessed by relating heart rate (HR) fluctuations to blood pressure (BP) fluctuations. Change in BRS after salmeterol inhalation is expressed in terms of milliseconds per millimeters of mercury (ms/mmHg). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0 before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the specified time points were assessed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
ms/mmHg
  Change from Baseline to 2 hours, Week 0, n=31 | 0.1 (1.9)
  Change from Baseline to Week 4, n=29 | 0.2 (2.6)

20. Secondary Outcome: Change From Baseline in Spontaneous Baroreflex Sensitivity (BRS) at 2 Hours (Week 0) and at Week 4 (ITT-MSNA Population)
Description: as for outcome 19
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT-MSNA Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 17
ms/mmHg
  Change from Baseline to 2 hours, Week 0 | 0.28 (2.2)
  Change from Baseline to Week 4 | 0.44 (3.2)

21. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at 2 Hours (Week 0) and at Week 4 (ITT Population)
Description: Pulmonary function was measured by FEV1, defined as the volume of air that which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Change in FEV1 after salmeterol inhalation is expressed in terms of liters (L). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
L
  Change from Baseline to 2 hours, Week 0, n=32 | -0.04 (0.23)
  Change from Baseline to Week 4, n=31 | -0.04 (0.21)

22. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at 2 Hours (Week 0) and at Week 4 (ITT-MSNA Population)
Description: as for outcome 21
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT-MSNA Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 18
L
  Change from Baseline to 2 hours, Week 0 | -0.05 (0.26)
  Change from Baseline to Week 4 | -0.08 (0.21)

23. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure (BP) at 2 Hours (Week 0) and at Week 4
Description: Systolic and diastolic BP was manually measured. Change in BP after salmeterol inhalation is expressed in terms of millimeters of mercury (mmHg). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 31
mmHg
  Systolic: Change from Baseline to 2 hours, Week 0 | 3.6 (12.3)
  Systolic: Change from Baseline to Week 4 | 3.7 (15.7)
  Diastolic: Change from Baseline to 2 hours, Week 0 | 1.9 (6.7)
  Diastolic: Change from Baseline to Week 4 | 0.7 (6.8)

24. Secondary Outcome: Change From Baseline in Respiratory Rate at 2 Hours (Week 0) and at Week 4
Description: Respiratory rate is defined as the number of breaths taken within a set amount of time (typically within 60 seconds). Change in respiratory rate after salmeterol inhalation is expressed in terms of respiratory rate (breaths) per minute (min). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
breaths per minute
  Change from Baseline to 2 hours, Week 0, n=32 | -0.5 (1.6)
  Change from Baseline to Week 4, n=31 | -0.1 (2.6)

25. Secondary Outcome: Change From Baseline in Tidal Volume at 2 Hours (Week 0) and at Week 4
Description: Tidal volume is defined as the lung volume representing the normal volume of air displaced between normal inspiration and expiration when extra effort is not applied (normal value is approximately 500 milliliters or 7 milliliters per kilogram of body weight). Change in tidal volume after salmeterol inhalation is expressed in terms of milliliters (mL). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
mL
  Change from Baseline to 2 hours, Week 0, n=30 | 60.4 (118.0)
  Change from Baseline to Week 4, n=24 | 55.6 (183.7)

26. Secondary Outcome: Change From Baseline in Respiratory Minute Volume at 2 Hours (Week 0) and at Week 4
Description: Respiratory minute volume is defined as the volume of gas inhaled (inhaled minute volume) or exhaled (exhaled minute volume) from a person's lungs per minute. Change in respiratory minute volume after salmeterol inhalation is expressed in terms of milliliters per minute (mL/min). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
mL/min
  Change from Baseline to 2 hours, Week 0, n=30 | 572.0 (1529.7)
  Change from Baseline to Week 4, n=24 | 671.4 (2963.3)

27. Secondary Outcome: Change From Baseline in Catecholamines (Plasma Norepinephrine) at 2 Hours (Week 0) and at Week 4
Description: Catecholamines are important neurotransmitters in the central nervous system and play a crucial role in the autonomic regulation of many homeostatic functions. Change in catecholamines (plasma norepinephrine) after salmeterol inhalation is expressed in terms of nanogramms per liter (ng/L). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
ng/L
  Change from Baseline to 2 hours, Week 0, n=26 | -42.4 (103)
  Change from Baseline to Week 4, n=29 | -5.7 (133)

28. Secondary Outcome: Change From Baseline in Catecholamines (Plasma Epinephrine) at 2 Hours (Week 0) and at Week 4
Description: Catecholamines are important neurotransmitters in the central nervous system and play a crucial role in the autonomic regulation of many homeostatic functions. Change in catecholamines (plasma epinephrine) after salmeterol inhalation is expressed in terms of nanograms per milliliter (ng/mL). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
ng/mL
  Change from Baseline to 2 hours, Week 0, n=26 | 6.7 (12.7)
  Change from Baseline to Week 4, n=29 | -0.3 (10.4)

29. Secondary Outcome: Change From Baseline in Catecholamines (Brain Natriuretic Peptide [BNP]) at 2 Hours (Week 0) and at Week 4
Description: Catecholamines are important neurotransmitters in the central nervous system and play a crucial role in the autonomic regulation of many homeostatic functions. Change in catecholamines (BNP) after salmeterol inhalation is expressed in terms of picograms per milliliter (pg/mL). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 27
pg/mL
  Change from Baseline to 2 hours, Week 0 | 2.4 (7.0)
  Change from Baseline to Week 4 | -6.1 (28.5)

30. Secondary Outcome: Change From Baseline in Oxygen Saturation Measured Via Pulse Oxymetry (SpO2) at 2 Hours (Week 0) and at Week 4
Description: Oxygen saturation measures the capacity of blood to transport oxygen to other parts of the body. Oxygen binds to hemoglobin in red blood cells when moving through the lungs. A pulse oximeter uses two frequencies of light (red and infrared) to determine the percentage of hemoglobin in the blood that is saturated with oxygen. The percentage is called blood oxygen saturation, or SpO2. Change in SpO2 after salmeterol inhalation is expressed in terms of percent. Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: Safety Population: all participants included in the study who received at least one dose of study medication. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
percent
  Change from Baseline to 2 hours, Week 0, n=32 | -0.2 (1.1)
  Change from Baseline to Week 4, n=31 | -0.5 (2.0)

31. Secondary Outcome: Change From Baseline in Transcutaneous Carbon Dioxide (tCO2) at 2 Hours (Week 0) and at Week 4
Description: Transcutaneous carbon dioxide monitoring is a noninvasive way of continuously measuring the tension of these gases in the skin. This methodology provides a continuous noninvasive estimation of the arterial CO2 value. Change in tCO2 after salmeterol inhalation is expressed in terms of millimeters of mercury (mmHg). Change from Baseline was calculated as the value at 2 hours (Week 0 [Visit 1, after salmeterol inhalation]) and the value at Week 4 (Visit 2, after salmeterol inhalation) minus the value at Baseline (Week 0, before any inhalation).
Time Frame: Baseline, 2 hours (Week 0), and Week 4
Population: Safety Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
mmHg
  Change from Baseline to 2 hours, Week 0, n=32 | -0.94 (2.19)
  Change from Baseline to Week 4, n=31 | -0.82 (4.17)

32. Secondary Outcome: Lung Function (Forced Vital Capacity [FVC], Functional Residual Capacity [FRC; Body and Helium], Total Lung Capacity [TLC], and Residual Volume [RV]) at Baseline (Week 0) and at Week 4
Description: FVC is defined as the volume of air that can be forcibly blown out from the lungs after a full inspiration. FRC is defined as the volume of air present in the lungs, specifically the parenchyma tissues, at the end of a passive expiration. TLC is defined as the maximum volume to which the lungs can be expanded with the greatest possible inspiratory effort; it is equal to VC plus the RV and is approximately 5800 milliliters. RV is defined as the amount of gas remaining in the lungs at the end of a maximal exhalation. All parameters describing lung function are expressed in terms of liters (L). Lung function (FVC, FRC [body and helium], TLC, and RV) was evaluated at Baseline (Week 0, [Visit 1, before any inhalation]) and at Week 4 (Visit 2, after salmeterol inhalation).
Time Frame: Baseline and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
L
  FVC at Baseline, Week 0, n=32 | 2.60 (0.7)
  FVC at Week 4, n=31 | 2.64 (0.7)
  FRC (body) at Baseline, Week 0, n=32 | 4.65 (1.3)
  FRC (body) at Week 4, n=27 | 3.67 (1.8)
  FRC (helium) at Baseline, Week 0, n=24 | 3.64 (1.0)
  FRC (helium) at Week 4, n=24 | 3.38 (0.8)
  TLC at Baseline, Week 0, n=32 | 6.61 (1.4)
  TLC at Week 4, n=27 | 5.67 (1.8)
  RV at Baseline, Week 0, n=32 | 3.90 (1.3)
  RV at Week 4, n=27 | 2.90 (1.8)

33. Secondary Outcome: Number of Participants With Diastolic Dysfunction on Echocardiography at Baseline (Week 0) and at Week 4
Description: Diastolic dysfunction refers to the decline in performance of one (usually the left ventricle) or both (left and right) ventricles during diastole. The number of participants with diastolic dysfunction on echocardiography was evaluated at Baseline (Week 0, [Visit 1, before any inhalation]) and at Week 4 (Visit 2, after salmeterol inhalation).
Time Frame: Baseline and Week 4
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Number; unit: participants
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
participants
  Baseline: Diastolic dysfunction: Yes, n=32 | 3
  Baseline: Diastolic dysfunction: No, n=32 | 29
  Week 4: Diastolic dysfunction: Yes, n=31 | 5
  Week 4: Diastolic dysfunction: No, n=31 | 26

34. Secondary Outcome: Arterial Stiffness at Baseline (Week 0) and at Week 4
Description: Arterial stiffness occurs as a consequence of age and arteriosclerosis. Carotid-femoral pulse wave velocity (PWV), a measure of arterial stiffness, is determined from the time taken for the arterial pulse to propagate from the carotid to the femoral artery. PWV was evaluated in terms of meters per second (m/s). PWV after salmeterol inhalation at Baseline (Week 0, [Visit 1, before any inhalation]) and at Week 4 (Visit 2, after inhalation of salmeterol) was assessed.
Time Frame: Baseline and Week 4
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Salmeterol 50 µg BID
Number analyzed (Participants) | 32
m/s
  PWV at Baseline, Week 0, n=30 | 9.2 (2.1)
  PWV at Week 4, n=29 | 8.8 (2.2)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study medication to the end of treatment (up to 37 days/average of 28.2 days)
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of trial medication during the treatment period.
Arm/Group | Salmeterol 50 µg BID
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 19/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Salmeterol 50 µg BID (N=32)
Palpitations (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Swollen tongue (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.